CLINICAL TRIAL: NCT03071575
Title: Assessing Immunogenicity of Measles-Rubella Vaccine at 6 and 9 Months of Age
Brief Title: Measles-Rubella Vaccine Immunogenicity at 6 and 9 Months of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Ministry of Health and Family Welfare, Bangladesh (Unknown)
Responsible Party: Principal Investigator, Jennifer Knapp, Epidemiologist, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC
Record Dates: First submitted 2017-02-21; First posted 2017-03-07 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Measles; Rubella; Rubella Syndrome, Congenital
Keywords: measles; rubella; immunogenicity; congenital rubella syndrome; measles-rubella vaccine
MeSH Terms: conditions — Measles; Rubella; Rubella Syndrome, Congenital | interventions — Aging

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: early dose (Experimental): Infants receive a measles-rubella vaccine at 6 and 9 months. Infants receive a standard dose according to the vaccine package insert each time. (Mothers receive no intervention.)
  Interventions: Biological: Measles-rubella (MR) vaccine at 6 months of age; Biological: Measles-rubella (MR) vaccine at 9 months of age
- Group B: standard dose (Active Comparator): Infants receive a measles-rubella vaccine at 9 months only. Infants receive a standard dose according to the vaccine package insert. (Mothers receive no intervention.)
  Interventions: Biological: Measles-rubella (MR) vaccine at 9 months of age

INTERVENTIONS:
Biological: Measles-rubella (MR) vaccine at 6 months of age — Infants receive a standard dose according to the vaccine package insert. (Mothers receive no intervention.)
  Other Names: Early dose
  Arms: Group A: early dose
Biological: Measles-rubella (MR) vaccine at 9 months of age — Infants receive a standard dose according to the vaccine package insert. (Mothers receive no intervention.)
  Other Names: Standard dose

SUMMARY:
This is an open-label, randomized, 2-arm clinical trial in healthy infants in Bangladesh. The primary purpose of the study is to assess the immunogenicity of measles-rubella (MR) vaccine when delivered at 6 months. In addition, the study will establish the equality of MR vaccine seroconversion administered at 9 months following administration of an earlier MR vaccine dose at 6 months of age compared to MR vaccine dose administered at 9 months without previous MR vaccination. This study will also provide additional data on safety and tolerance of MR vaccine given at 6 months, and impact of maternal antibodies on immunogenicity of MR vaccine at 6 months.

* Primary objectives:

  1. To assess immunogenicity of MR vaccine at 6 months of age
  2. To assess immunogenicity of MR vaccine at 9 months of age among children without prior measles and rubella vaccination, compared with MR vaccine immunogenicity among those who had a prior MR vaccination at 6 months of age
* Secondary objectives

  1. To assess the frequency of adverse reactions following administration of MR vaccine at 6 months
  2. To compare the immunogenicity of the MR vaccine first dose administered at 6 months vs at 9 months.
  3. To assess the proportion of mothers with undetectable, detectable and protective levels of measles and rubella antibodies
  4. To determine the extent of variation in measles antibodies in women of child bearing age in a population with a long standing measles vaccination program
  5. To determine the extent of variation in rubella antibodies in women of child bearing age in a population where rubella vaccine have been recently introduced
  6. To determine if variation in antibody levels in infants at 6 months is predominately explained by variation in starting antibody levels in the mother in this population
  7. To estimate the half-life of decay of measles and rubella antibodies in infants

DETAILED DESCRIPTION:
In countries with low levels of circulating measles virus, and lower risk for measles infection, measles containing vaccine first dose (MCV1) is recommended at 12 months of age. In countries with high risk for measles, MCV1 is recommended at 9 months. In the past decade, many countries have been experiencing measles outbreaks with a high proportion of cases among infants < 9 months of age, below the recommended age of routine MCV1.

Recent publications suggest that this may be due to the fact that the majority of infants now are born to mothers with vaccine induced immunity to measles, and who lose maternal antibodies much earlier, by age of 4-6 months. For example, in a measles outbreak in Malawi in 2010, 14% (17,858) of the estimated 134,000 cases occurred in children 0-8 months. In 2013, in a measles outbreak in Sri Lanka approximately 34% of measles cases were in children 6-12 months of age. Furthermore, in 2013 Jordan experienced a large measles outbreak with high proportion of young infants affected (6-9 months). WHO measles outbreak response guidelines recommend vaccinating children as young as 6 months during outbreaks. As an example, in response to a measles outbreak, Sri Lanka and Jordan conducted outbreak response immunization (ORI) that included infants 6 months of age despite the limited evidence on immunogenicity of MR vaccine at that age.

Some researchers suggest that routine MCV should be given before age of 9 months based on published data showing that infants born to mothers with vaccine induced measles immunity are born with lower concentration of maternal measles antibodies (MMA) and lose protection against measles infection at an earlier age. Measles vaccine immunogenicity depends on several factors, including presence of maternal measles antibodies (i.e., passively acquired measles antibodies may neutralize vaccine virus before a complete immune response develops resulting in primary vaccine failure.), maturity of immune system of the vaccine recipient, and strain of the measles vaccine used. So any decisions to alter the age of MCV1 dose should balance the potential risk of primary vaccine failure against the risk of measles infection and measles related complications, including death. Immunogenicity of measles vaccine given at 6 months is well studied; however, data on immunogenicity of combined MR vaccine administered at 6 months and its impact on MR vaccine effectiveness given at 9 months, is limited.

Because the number of infants born to mothers with vaccine induced immunity has been steadily increasing and most countries will be using MR vaccine routinely in the Expanded Program of Immunization (EPI), it is timely to conduct a study to assess immunogenicity of MR vaccine given at 6 months and its impact on a subsequent 9 month MR dose. The first dose of MCV given at 6 months is frequently referred to as MCV-0, indicating that two subsequent doses are needed to attain population seroprotection levels necessary to stop endemic transmission of the measles virus.

To improve the accuracy of interpretation of study results blood samples of mothers of enrolled infants will be tested for measles and rubella antibodies. This will also enable us to determine the proportion of mothers with undetectable, detectable and protective levels of antibodies, and to assess the relationship between the level of antibodies in mothers and their infants' maternal antibodies.

This study will be conducted in a single site in rural Bangladesh at Matlab. Matlab is a major rural field site for icddr,b, where for the past 50 years continuous health and demographic information was collected on >200,000 population.

From 2007 to 2010, icddr,b, the Ministry of Health (MOH) in collaboration with other international organizations conducted several randomized vaccine effectiveness studies.

This study will be an open-label, randomized, 2-arm clinical trial. 620 children will be enrolled and randomized at 6 months of age to one of two study arms. The primary objectives of this study are to assess the immunogenicity of MR vaccine at 6 months, and assess equality of MR vaccine seroconversion administered at 9 months following administration of an earlier MR vaccine dose at 6 months of age compared with MR vaccine dose administered at 9 months only without previous MR vaccination. The study will enroll generally healthy 6 month old infants living in Matlab and who have never received an MR vaccine dose and have no history of measles or rubella. Participants will be followed to 11 months of age.

Infants in this study will be randomly assigned to one of two arms. Infants in Study Arm A will receive MR vaccine at 6 months of age (at enrolment) and at 9 months. Infants in Study arm B will receive MR vaccine only at 9 months.

Blood specimens will be collected from all infants at 6, 9 and 11 months of age. The 6 month sample is a pre-vaccination sample and mainly will be used to determine maternal antibody levels. For arm A, the sample collected at 9 months before the second MR dose will be used to assess antibody levels after the first MR dose at 6 months of age. For study Arm B, the 9 month sample will be used to assess measles and rubella antibody decay rate. The sample collected at 11 months will be used to assess immune response to either a two dose or a one dose schedule (arms A and B, respectively).

ELIGIBILITY:
Age is based on the age of the infant.

Inclusion Criteria: INFANTS:

* Healthy infants at 6 months (180 days, +/- 7 days) of age
* A parent or guardian that consents for participation in the full length of the study
* A parent or guardian that is able to understand and comply with planned study procedures

Inclusion criteria: MOTHERS:

* Mothers of infants that meet inclusion criteria.
* ≥18 years of age
* Mothers who consent to participate in the full length of the study

Exclusion Criteria: INFANTS:

* Family that is unable to participate in the full length of the study
* A diagnosis or suspicion of immunodeficiency disorder either in the infant or mother
* A diagnosis or suspicion of bleeding disorder that would contraindicate parenteral administration of MR vaccine or collection of blood by venipuncture
* Acute infection or illness at the time of enrollment (6 months) that would require infant's admission to a hospital
* Receipt of any measles or rubella containing vaccine prior to enrolment (i.e., before age 6 months) outside of study based upon documentation or parental recall
* Known history of laboratory confirmed measles or rubella infection
* A diagnosis of rubella infection in mother during pregnancy
* A diagnosis of congenital rubella syndrome in infant
* Known allergy/sensitivity or reaction to measles-rubella containing vaccine or contents of measles-rubella containing vaccine
* Persons with a history of an anaphylactic reaction to any components of the vaccine
* Infants from premature births (<37 weeks of gestation)

Exclusion criteria: MOTHERS:

* Refuses to give blood samples. (If the mother agrees for her child to participate in the study, but refuses to give a blood samples herself or blood samples cannot be obtained, the child will still be enrolled.)
* A diagnosis or suspicion of immunodeficiency disorder
* A diagnosis or suspicion of bleeding disorder that would contraindicate collection of blood by venipuncture

Temporary exclusion: INFANTS:

* Acute febrile illness (≥38°C) at the time of enrollment
* Family will be requested to bring back the child 1-2 days later or when child feels better.

Ages: 173 Days to 187 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 637 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-03-18 (Actual); Study Completion 2018-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Zaman, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B, Chāndpur, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sayi TS, Sharapov UM, Matson Z, Coughlin MM, Crooke SN, An Q, Knapp JK, Aziz AB, Yunus M, Haque W, Rana S, Khan MAF, Alexander JP, Kretsinger K, Rota PA, Zaman K, Anand A. Immunogenicity and safety of a measles and rubella-containing vaccine at age 6 and 9 months in Bangladesh: an open-label, randomised trial. Lancet Child Adolesc Health. 2025 May;9(5):306-314. doi: 10.1016/S2352-4642(25)00090-2. Epub 2025 Mar 31. PMID 40179934

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 637 mother/infant dyads assessed for eligibility, 620 met inclusion criteria and were randomized to either Group A or Group B.
Period: Overall Study
Arm/Group | Group A: Early Dose | Group B: Standard Dose
Started | 312 | 308
Completed (This table presents information about whether the maternal infant/dyad completed all required study check-ins. Additional exclusions occurred at the analysis stage, where key blood specimens, while collected, were insufficient to provide the necessary information for analysis.) | 303 | 294 (One infant died after enrollment/randomization and before the second study time point. The infant did not receive the intervention and did not complete this study and was excluded from analysis (except reported in the adverse events all-cause mortality section).)
Not Completed | 9 | 14
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 5 | 11
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Population: Group A and group B, each had 2 participants without laboratory results and were removed from the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Early Dose | Group B: Standard Dose | Total
Number analyzed (Participants) | 301 | 292 | 593
Age, Continuous [Mean (Standard Deviation); unit: days] — Age of Infant
  days | 179.8 (3.3) | 179.5 (3.3) | 179.7 (3.3)
Age, Continuous [Mean (Standard Deviation); unit: years] — Maternal age at enrollment
  years | 26.5 (5.4) | 26.4 (5.6) | 26.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of the infant, the mothers of the infants were female.
  Participants
    Female | 156 | 146 | 302
    Male | 145 | 146 | 291
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Stunting present [Count of Participants; unit: Participants] | 29 | 35 | 64
Wasting present [Count of Participants; unit: Participants] | 15 | 12 | 27
Measles seropositivity (Infants) [Count of Participants; unit: Participants] | 10 | 6 | 16
Rubella seropositivity (Infants) [Count of Participants; unit: Participants] | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent of Infants Who Were Seropositive After Immunization at 6 Months (Assessed at 9-month Visit)
Description: # seropositive infants at 9 months/ # of infants in the arm Measles neutralizing antibody titers as measured by plaque reduction neutralization assay is defined as seropositive at ≥ 120 mIU/mL.
  Rubella antibody titers as measured by ELISA are considered seropositive at >10 IU/mL. Abbreviations mIU =milli-International unit; IU International units; mL milliliter
Time Frame: Infant antibody titer at 9 months.
Population: This is an analysis of Group A infants only, as Group B infants did not receive a vaccine at 6 months. (No mothers were vaccinated in this study)
Measure: Number (95% Confidence Interval); unit: percentage of infants
Groups:
- Group A:: Infants receive a measles-rubella vaccine at 6 and 9 months. Infants receive a standard dose according to the vaccine package insert each time. (Mothers receive no intervention.)
Arm/Group | Group A:
Number analyzed (Participants) | 301
percentage of infants
  Measles | 94 [90 to 96]
  Rubella | 94 [91 to 96]

2. Primary Outcome: Percent of Infants Who Were Seropositive After Immunization at 9 Months (Assessed at 11-month Visit)
Description: # seropositive at 11 months of age/ # of infants in the arm * 100 Measles neutralizing antibody titers as measured by plaque reduction neutralization assay is defined as seropositive at ≥ 120 mIU/mL.
  Rubella antibody titers as measured by ELISA are considered seropositive at >10 IU/mL. Abbreviations mIU =milli-International unit; IU International units; mL milliliter
Time Frame: Infant antibody titer at 11 months.
Population: Infants only, no mothers were vaccinated as part of this study.
Measure: Number (95% Confidence Interval); unit: percentage of infants
Arm/Group | Group A: Early Dose | Group B: Standard Dose
Number analyzed (Participants) | 301 | 292
percentage of infants
  Measles | 99 [97 to 100] | 100 [98 to 100]
  Rubella | 99 [96 to 100] | 100 [98 to 100]

3. Secondary Outcome: Adverse Effects Following Immunization (AEFI) at the Age of 6 Months
Description: To assess the frequency of adverse reactions following administration of MR vaccine at the age of 6 months. There were multiple assessment timeframes relative to the first immunization. 30 minutes direct observation at the clinic site and 48-hour follow-up visit by study staff at the home.
Time Frame: 0-30 minutes; 48-hour visit.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Early Dose
Number analyzed (Participants) | 301
Participants
  Redness at the injection site (in 30 minutes) | 3
  Redness at the injection site (0.5 to 48 hours) | 0
  Fever (in 48 hours) | 7
  Cough, coryza, sneezing, or cold (in 48 hours) | 5
  Rash (in 48 hours) | 1
  No Vaccine Reaction reported (in 48 hours) | 285

4. Secondary Outcome: Immunogenicity at 9 Months - Measles
Description: The average antibody levels of infants who seroconverted or responded to the measles component of the vaccine. This measures the number of antibodies against the measles virus per volume of blood. A larger number means more antibodies are present and suggests a better ability to detect and prevent infection by the measles virus.
Time Frame: At 9 months and 11 months of age
Population: This value is only available for infants who seroconverted and produced measurable IgG antibodies against measles.
Measure: Median (Inter-Quartile Range); unit: mIU/mL
Arm/Group | Group A: Early Dose | Group B: Standard Dose
Number analyzed (Participants) | 297 | 291
mIU/mL
  IgG at 9 months of age: number analyzed (Participants) | 282 | 0
  IgG at 9 months of age | 914 [584 to 1353] |
  IgG at 11 months of age | 1453 [1057 to 2094] | 1311 [881 to 1976]

5. Secondary Outcome: Immunogenicity at 9 Months - Rubella
Description: The average antibody levels of infants who seroconverted or responded to the rubella component of the vaccine. This measures the number of antibodies against the rubella virus per volume of blood. A larger number means more antibodies are present and suggests a better ability to detect and prevent infection by the rubella virus.
Time Frame: At 9 months and 11 months of age
Population: This value is only available for infants who seroconverted and produced measurable IgG antibodies against rubella.
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | Group A: Early Dose | Group B: Standard Dose
Number analyzed (Participants) | 297 | 291
IU/mL
  IgG at 9 months of age: number analyzed (Participants) | 283 | 0
  IgG at 9 months of age | 102 [59 to 166] |
  IgG at 11 months of age | 94 [60 to 137] | 155 [91 to 228]

6. Secondary Outcome: Measles and Rubella Titers of Enrolled Mothers
Description: To assess the distribution of mothers with undetectable, detectable and protective levels of measles and rubella immunoglobulin G (IgG) antibodies
Time Frame: Baseline enrollment (when infant was 6 months of age)
Measure: Count of Participants; unit: Participants
Groups:
- Group A: Mothers: Infants who receive a measles-rubella vaccine at 6 and 9 months. Infants receive a standard dose according to the vaccine package insert each time. (Mothers receive no intervention.)
- Group B: Mothers: Infants receive a measles-rubella vaccine at 9 months only. Infants receive a standard dose according to the vaccine package insert. (Mothers receive no intervention.)
Arm/Group | Group A: Mothers | Group B: Mothers
Number analyzed (Participants) | 301 | 292
Participants
  Measles IgG (Undetectable: <4mIU/mL; Protective: at least 153 mIU/mL): Undetectable | 0 | 0
  Measles IgG (Undetectable: <4mIU/mL; Protective: at least 153 mIU/mL): Detectable | 46 | 37
  Measles IgG (Undetectable: <4mIU/mL; Protective: at least 153 mIU/mL): Protective | 255 | 255
  Rubella IgG (Undetectable: <0.08 IU/mL; Protective: at least 9·36 IU/mL): Undetectable | 0 | 0
  Rubella IgG (Undetectable: <0.08 IU/mL; Protective: at least 9·36 IU/mL): Detectable | 52 | 53
  Rubella IgG (Undetectable: <0.08 IU/mL; Protective: at least 9·36 IU/mL): Protective | 249 | 239

7. Secondary Outcome: Pearson Correlation Coefficient of Infant Measles and Rubella Antibody Levels at 6, 9, and 11 Months of Age Compared to Maternal Antibody Levels at Baseline (a Proxy for Infant Antibody Levels at Birth).
Description: Pearson correlation coefficient, by arm at each study timepoint. It quantifies the linear relationship between two sets of variables; we compare the infant antibody levels (y axis) to that of the mother at baseline (x-axis), a proxy for infant antibody levels at birth. This is usually presented as a scatter plot. A coefficient approaching 1 or -1 indicates a strong correlation, while a coefficient near zero indicates no correlation.
Time Frame: baseline (6 months infant age); 2nd blood draw (9 months of age) and 3rd blood draw (at 11 months of age)
Population: This looks at the variation in the infant's antibody response overtime compared to a maternal baseline (a proxy for the infant's antibody level at birth).
Measure: Number; unit: Pearson correlation coefficient (r)
Groups:
- Group A: Early Dose: Infants who receive a measles-rubella vaccine at 6 and 9 months. Infants receive a standard dose according to the vaccine package insert each time. (Mothers receive no intervention.)
Arm/Group | Group A: Early Dose | Group B: Standard Dose
Number analyzed (Participants) | 301 | 292
Pearson correlation coefficient (r)
  Measles baseline (6 months) | 0.72 | 0.66
  Measles (9 months) | -0.26 | 0.32
  Measles (11 months) | -0.03 | 0.02
  Rubella baseline (6 months) | 0.74 | 0.74
  Rubella (9 months) | -0.27 | 0.51
  Rubella (11 months) | -0.19 | -0.11

8. Secondary Outcome: Half-life and Decay of Maternal Measles and Rubella Antibodies.
Description: To estimate the half-life of decay of maternal measles and rubella antibodies in infants
Time Frame: Day 1 to day 84
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Infants were assessed 0-30 minutes following immunization at the clinic, and parents were queried for adverse events at each subsequent study visit, up to 5 months in total duration. Arm A also received a safety monitoring visit at home 48 hours after immunization following the 6-month visit.
Description: Only infants were assessed for adverse events. Additional exclusions are based on patient flow (eg. loss to follow-up, withdrawal of consent).
Groups:
- Group A: Early Dose: Infants receive a measles-rubella vaccine at 6 and 9 months. Infants receive a standard dose according to the vaccine package insert each time. (Mothers receive no intervention and were not monitored for any adverse events.) After the 6-month vaccination, these participants also received a 48-hour safety monitoring visit at their home.
- Group B: Standard Dose: Infants receive a measles-rubella vaccine at 9 months only. Infants receive a standard dose according to the vaccine package insert. (Mothers receive no intervention and were not monitored for any adverse events.) [Note: The infant death happened before any vaccine was given; and was excluded from study analyses.]
Arm/Group | Group A: Early Dose | Group B: Standard Dose
All-Cause Mortality (participants affected / at risk) | 0/312 | 1/308
Serious Adverse Events (participants affected / at risk) | 10/312 | 7/308
Other Adverse Events (participants affected / at risk) | 38/312 | 31/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Early Dose (N=312) | Group B: Standard Dose (N=308)
Hospitalization: Respiratory Infections (Infections and infestations) | 5 (6) | 4 (4)
Surgical procedure (Surgical and medical procedures) | 1 (1) | 1 (1)
Hospitalization: other (Infections and infestations) | 6 (7) | 2 (2) — Includes: diarrhea, urinary and skin infections.
Anaphylaxis (Immune system disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Early Dose (N=312) | Group B: Standard Dose (N=308)
Respiratory Infection (Infections and infestations) | 29 (30) | 25 (26)
Diarrhea (Infections and infestations) | 7 (7) | 5 (5)
Varicella (Chicken Pox) (Infections and infestations) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT03071575/Prot_SAP_ICF_000.pdf